CLINICAL TRIAL: NCT07252492
Title: Evaluation of Performances, Clinical Benefits and Safety of the 'Audiocap' Connected Hearing Rehabilitation Device for Improving Audibility in Hearing-impaired People in the Context of CE Marking
Brief Title: Evaluation of Performances, Clinical Benefits and Safety of the 'Audiocap' Connected Hearing Rehabilitation Device for Improving Audibility in Hearing-impaired People in the Context of CE Marking - AUDIOCAP-2
Acronym: AUDIOCAP-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Archean Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-A01026-43
Record Dates: First submitted 2025-09-11; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Adult-Onset; Hearing Aid
Keywords: Aides auditives; Prothèses auditives; Perte auditive; Appareillage audition; Adulte audition
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: First period of one month: Double blinded randomized placebo-controlled trial (Placebo/group A versus Audiocap standard mode/ group B).
  Interventional Arm: Audiocap connected hearing aid in a standard interplay path.
  Control Arm: Audiocap connected hearing aid with a 'NONE' setting (flat frequency response for the patient (equivalent to not wearing hearing aid) in a standard interplay path.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Active Comparator): First period of one month: Audiocap connected hearing aid in a standard interplay path.
  Interventions: Device: Audiocap connected hearing aid
- Control Arm (Placebo Comparator): First period of one month: Audiocap connected hearing aid with a 'NONE' setting (flat frequency response for the patient (equivalent to not wearing hearing aid) in a standard interplay path.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Audiocap connected hearing aid — The hearing aids will be used in a standard mode, that is, without the possibility of remote adjustment (remote interplay path).
  Arms: Interventional Arm
Device: Placebo — Audiocap connected hearing aid with a 'NONE' setting (flat frequency response for the patient (equivalent to not wearing hearing aid) in a standard interplay path.
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is the evaluation of performances, clinical benefits and safety of the 'Audiocap' connected hearing rehabilitation device for improving audibility in hearing-impaired people.

The main question it aims to answer is to demonstrate, after one month's use of the Audiocap connected hearing aid, that the audiological gain for the patient is better than with a placebo hearing aid.

Placebo hearing aid is a Audiocap connected hearing aid with a 'NONE' setting (flat frequency response for the patient (equivalent to not wearing hearing aid).

Participants will be first-time hearing aid users, eligible for hearing aid fitting, and adults according to French legislation (18 years and older).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting one or more of the following criteria: a.Subject with mild to moderate hearing loss (20dB to 50dB average at 500, 1000, 2000, and 4000 Hz) in the better ear according to WHO standards, / b. Subject with a speech reception threshold (SRT) in quiet exceeding 30dB, corresponding to the minimum speech level required to achieve 50% recognition in silence (HAS eligibility criteria for hearing aid reimbursement), / c. Subject with significant degradation of speech intelligibility in noise, defined as a speech-to-noise ratio (SNR) deviation greater than 3dB compared to normative reference values (HAS eligibility criteria for hearing aid reimbursement), / d.Subject with high-frequency hearing loss greater than 30dB from 2000 Hz onwards, associated with a speech reception threshold exceeding 30dB in quiet and/or a significantly degraded speech intelligibility in noise (HAS eligibility criteria for hearing aid reimbursement).
2. Subjects eligible for first hearing aid.
3. Subjects over 18 years of age. French-speaking subjects.

5. Subjects affiliated with a social security scheme. 6. Subjects who are not subject to another medical option, without external pathology and excluding implants.

7. Subjects who have signed an informed consent. 8. Subjects available for the study.

Exclusion Criteria:

1. Subject deprived of his/her liberty by a judicial or administrative decision
2. Subject with severe psychiatric disorder
3. Subject admitted to a health or social care establishment
4. Subject not able to give consent
5. Adults under guardianship or trusteeship.
6. Subjects with disabling tinnitus that are not suitable for adaptation (THI>56).
7. Subjects eligible for a cochlear implant.
8. Subjects not able to participate in the study according to the investigator.
9. Subjects with acute and chronic suppurative otitis media, congenital ear atresia, or any type of ear discharge.
10. Subjects with congenital atresia of external ear or deformity of any part of the ear canal.
11. Subjects with deafness that is unstable and with a degree of hearing loss often fluctuating.
12. Subjects with persistent headaches, dizziness, earaches, or other symptoms that are not suitable for adaptation.
13. Subjects with sudden onset of hearing loss within the past 3 months, rapid progressive deafness, unilateral hearing loss or other acute ear disease.
14. Subjects with effusion (secretions/ discharge) in the ear and/or frequent purulence (pus).
15. Subjects with central deafness (central nervous system) or non-organic deafness.
16. Subjects with acute otitis extrema and tympanitis.
17. Subjects who are allergic to materials of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the Audiocap connected hearing aid will be measured by the improvement of at least one of the following three audiological gain criteria. | After one month of hearing aid use (Month 1)
  The effectiveness of the Audiocap connected hearing aid will be measured by the improvement of at least one of the following three audiological gain criteria:
  1. Mean tonal gain of 10 dB (mean 500 / 1000 / 2000 / 4000 Hz).
  2. Minimum vocal prosthetic gain of 7 dB (dissyllabic words).
  3. Improvement in speech in noise of at least 2 dB SNR (FrMatrix test).
  Clarification: The primary endpoint measures the audiological gain in decibels (dB) through standard audiometric tests. Three non-cumulative possibilities (i.e., at least one of the three improvements) are defined: depending on the patient's hearing loss, the improvement is not expressed in the same way.

SECONDARY OUTCOMES:
Measurement of quality of life using the SSQi15 questionnaire | After one month (Month 1) and at the end of follow-up (Month 3 and Month 4)
  Quality of life will be assessed using questionnaires SSQi15.
  The SSQ-15 (Speech, Spatial, and Qualities of Hearing Scale, 15-item version) is a questionnaire that evaluates real-life hearing situations related to speech understanding, spatial hearing, and perceived qualities of hearing.
Measurement of quality of life using the COSI questionnaire | After one month of using (Month 1) and at the end of the follow up (Month 3 and Month 4)
  The Client Oriented Scale of Improvement (COSI) is a clinical tool developed by the National Acoustic Laboratories to assess hearing aid outcomes. Patients identify up to five specific listening situations they wish to improve. After a period of use, they rate the perceived improvement and their final ability to hear in each situation.
Treatment preference (Likert) | After one month (Month 1) and at the end of the patient's follow-up (Month 3 and Month 4)
  The subject will be asked to indicate their preference between not using a hearing aid and using a hearing aid on a scale from 0 to 10.
Reduction of the time required to attain adaptation to the hearing aid (remote interplay path) | After one month (Month 1) and at the end of follow-up (Month 3 and Month 4)
  The advantage of the remote interplay path is assessed through:
  2.a.1. If necessary for the patient, number of adjustments requested and/or number of positive responses to requests from the application to adjust the setting compared with the standard mode,
  2.a.2. The number of adjustments requested in the remote interplay path during the first month is higher than the last month,
  2.a.3. Comparison of the time interval between the last setting remote requested and the standard last visit,
  2.a.4. Subjects in remote interplay path have an equal or better average wearing time than subject in standard interplay path,
  2.a.5. During the last month, subjects in remote interplay path don't use their previous setting and don't request a new one,
  2.a.6. During the last month, subjects in remote interplay path don't change significantly the global broadcast level of their hearing aid.
Remote interplay path empowers the subject to take control of and better manage their hearing loss. | After one month (Month 1) and at the end of follow-up (Month 3 and Month 4)
  Subject empowerment is assessed by the PAM-13 questionnaire.
Acceptability assessed by wearing time (data logging) | After one month (Month 1) and at the end of follow-up (Month 3 and Month 4)
  Acceptability assessed by wearing time (data logging).
Usability (Ergonomic questionnaire) | After one month of use (M1) and at the end of the follow up (M3 and M4).
  Usability assessed via the ergonomics questionnaire.
  The ergonomic questionnaire is specially custom to evaluate the medical device (clear information, typeface, visual presentation, design, use and use of each feature).
Safety of the device : reporting adverse events, serious adverse events and device deficiencies. | This endpoint is measured at each subject visit in the study (visit 2 (Day 15), visit 3 (Month 1), visit 4 (Day 45), visit 5 (Month 2) and visit 6 (Month 4)).
  Safety of the device : number of adverse events, serious adverse events and device deficiencies (in the context of CE marking)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Edouard Herriot, Lyon, France
  - Clinique de l'Oreille, Paris, France
  - Hôpital Lariboisière (APHP), Paris, France
  - Clinique Rive-Gauche, Toulouse, France

IPD SHARING:
Plan to Share IPD: No